CLINICAL TRIAL: NCT06634654
Title: An Artificial Intelligence-based Approach in Total Knee Arthroplasty: From Inflammatory Responses to Personalized Medicine
Acronym: AI-TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Umile Giuseppe Longo, Professor, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 179.24 CET2 cbm; PNRR-MCNT2-2023-12378237 (Other Grant/Funding Number: NextGenerationEU - Italian Ministry of Health PNRR (National Recovery and Resilience Plan): M6/C2_CALL 2023)
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: Artificial Intelligence; Total Knee Arthroplasty; Biomechanics; Orthopaedic surgery; Alarmins; Oxidative Stress; Cytokine; Knee Inflammation; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee; Lost to Follow-Up; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients who undergo total total knee arthroplasty (Experimental): The study population comprises 197 patients who require Total Knee Arthroplasty (TKA) due to symptomatic, end-stage knee osteoarthritis. Eligible participants are adults over the age of 18 years with functionally intact ligaments. Exclusion criteria include individuals with neurological or other conditions that affect their ability to participate in walking trials, those with inflammatory or infectious arthritis, previous significant knee surgeries such as articular fractures (excluding knee arthroscopy and meniscal surgery), and those with active tumors or who are pregnant. This population selection is aimed at assessing the efficacy of AI-integrated interventions in improving surgical outcomes and postoperative recovery in a homogeneous group affected by severe knee degeneration.
  Interventions: Procedure: Total Knee Arthroplasty; Diagnostic Test: Multifaceted diagnostic assessments; Behavioral: Follow-ups; Genetic: Genetic screening

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Total Knee Arthroplasty is performed using conventional surgical techniques.
Diagnostic Test: Multifaceted diagnostic assessments — Multifaceted diagnostic assessments involving genetic analysis, biomechanical data collection, radiographic imaging, and psychological evaluations.
Behavioral: Follow-ups — Postoperative follow-up includes behavioral interventions, such as lifestyle counseling and rehabilitation programs, tailored based on AI-driven insights into individual patient recovery profiles.
Genetic: Genetic screening — Genetic screening and analysis, including whole exome sequencing, are conducted to identify genetic markers that might influence the outcomes of knee arthroplasty. This data is utilized within AI models to predict patient-specific surgical outcomes and recovery processes.

SUMMARY:
Goal: The goal of this interventional study is to understand how multimodal preoperative data can predict outcomes after Total Knee Arthroplasty (TKA) and improve personalized medicine practices.

Participant Population: The study will enroll 197 patients suffering from symptomatic, end-stage knee osteoarthritis, who are above 18 years old and have functionally intact ligaments.

Main Questions:

* Can multimodal preoperative data, genetic predisposition, and psycho-behavioral characteristics predict outcomes after TKA?
* Can AI models effectively use this data to customize prostheses and surgical interventions, and predict patient outcomes? Comparison Group Information (If applicable): Not specified in the provided details.

Participant Tasks:

* Undergo TKA as per the normal clinical routine.
* Participate in pre- and post-surgical follow-ups including:
* Clinical-functional assessments.
* Administration of clinical scores.
* Collection of biological samples.
* Biomechanical analysis using a stereophotogrammetric system.
* Provide data for the comprehensive multimodal indexed database.

DETAILED DESCRIPTION:
Osteoarthritis is one of the most common causes of knee disorders, leading to pain, reduced mobility, and a decline in quality of life. Total knee arthroplasty (TKA) is one of the most established treatments for end-stage osteoarthritis. Despite advancements in surgical techniques, patient dissatisfaction remains high. After surgery, patients often experience swelling, pain, and difficulty with daily activities. Revision surgery is a major challenge, with aseptic loosening occurring in 15-20% of cases. Given the high disability rates and healthcare costs associated with TKA, optimizing patient care is crucial.

Artificial intelligence (AI) offers the potential to identify new care profiles. For the first time, AI can integrate multimodal datasets. This approach could lead to personalized treatment for knee osteoarthritis patients, in line with precision medicine principles. This study takes a multidisciplinary approach to better understand the causes of failure and dissatisfaction following TKA.

The primary aim of this study is is to create a multimodal database. This database will include structural, genetic, biomechanical, clinical, psychological, biological, stress-related, inflammatory, and demographic data. Using AI, the study aims to build predictive models for post-TKA outcomes. Insights from this research could improve patient management and lead to new therapeutic approaches.

Patients suffering from knee osteoarthritis at Fondazione Policlinico Universitario Campus Bio-Medico will be enrolled in this study if they meet the inclusion/exclusion criteria described above.

There are no risks for the patients recruited in the study. The total duration of the study is 5 years. The enrolment of patients will start on the 01/10/2024 and will last 12 months for each patient.

The Italian Ministry of Health and the Fondazione Policlinico Universitario Campus Bio-Medico supported this study.

The PI and also the main contact of this study is professor Umile Giuseppe Longo.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic, end-stage knee osteoarthritis
2. Ligaments functionally intact
3. Age: older than18 years old

Exclusion Criteria:

1. Neurological or other conditions affecting patients ability to join walking trials
2. Inflammatory or infectious arthritis
3. Previous articular fracture or knee surgery (excluding knee arthroscopy and meniscal surgery)
4. Active tumors or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Knee Society Score (KSS) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The KSS is a clinician-based assessment tool that evaluates both knee function and functional activities after knee replacement surgery.
  Minimum/Maximum Values: The KSS is divided into two parts: knee score and function score, with a combined score ranging from 0 to 100. Higher scores indicate a better outcome in terms of knee function and overall knee health.
Change From Baseline in Oxford Knee Score (OKS) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The OKS is used to assess pain and function in individuals undergoing knee surgery or experiencing knee osteoarthritis, focusing on the patient&amp;amp;amp;amp;amp;#39;s perspective.
  Minimum/Maximum Values: The OKS ranges from 0 to 48. Higher scores represent a better outcome, with less pain and better joint function.
Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The KOOS is widely used to evaluate short- and long-term patient-reported outcomes following knee injury or surgery.
  Minimum/Maximum Values: The KOOS assesses five dimensions: pain, symptoms, function in daily living, function in sports/recreation, and knee-related quality of life. Each subscale ranges from 0 to 100. Higher scores reflect a better outcome, indicating fewer symptoms and better function.
Change From Baseline in Forgotten Joint Score Short Form (FJS-12) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The FJS-12 measures how much a patient is aware of their joint in daily activities, particularly after joint replacement surgery, with higher scores reflecting greater joint integration.
  Minimum/Maximum Values: The FJS-12 ranges from 0 to 100. High scores indicate good outcomes

SECONDARY OUTCOMES:
Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The WOMAC is commonly used to evaluate pain, stiffness, and physical function in patients with osteoarthritis, particularly in the knee and hip.
  Minimum/Maximum Values: The WOMAC ranges from 0 to 96. High scores indicate best functional status level
Change from baseline in knee range of motion (ROM) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  Knee joint ROM (measured in degree) will be assessed during gait using a 3D motion capture system
Change from baseline in ground reaction forces at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  Ground reaction forces (measured in Newtons) during gait will be measured using force platforms synchronized with the 3D motion capture system
Change from baseline in center of pressure (CoP) at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The CoP (measured in meters) will be measured during gait using force platforms synchronized with the 3D motion capture system
Change from baseline in walking speed at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  Walking speed (measured in meters per seconds) will be extracted using force platforms synchronized with the 3D motion capture system
Change from baseline in cadence at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  Cadence (measured in steps per minute) will be assessed during gait using force platforms synchronized with the 3D motion capture system
Change from baseline in Step and Stride Length at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  Step and Stride length (measured in meters) will be evaluate during gait using force platforms synchronized with the 3D motion capture system
Change from baseline in osteoarthritis (OA) severity based on the Kellgren-Lawrence score at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The severity of OA will be assessed using the Kellgren-Lawrence global radiographic score. Changes in OA severity will be graded on a scale from 0 to 4, with 0 indicating no OA and 4 indicating severe OA
Change from baseline in joint alignment at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The changes in joint alignment (measured in degrees) will be evaluated using X-rays to determine any shifts in anatomical alignment post-surgery
Change from baseline in lateral distal femoral angle at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The lateral distal femoral angle (measured in degrees) will be measured using X-rays to assess the alignment of the femur
Change from baseline in medial proximal tibial angle at 12 months | Baseline (before surgery) and 12 months postoperatively
  The medial proximal tibial angle will be measured to evaluate tibial alignment. X-rays will be used to assess changes in medial proximal tibial angle (measured in degrees)
Change from baseline in joint line convergence angle at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The joint line convergence angle (measured in degrees) will be measured using X-rays to evaluate the alignment of the knee joint
Change from baseline in tibial slope at 12 months | Before surgery (Baseline) and at 12 months postoperatively
  The tibial slope (measured in degrees) will be assessed using X-rays to measure the posterior inclination of the tibial plateau
Change From Baseline in the fecal microbiota profiles at 12 months | Before surgery and at 12 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The ownership of the data is of the promoter and shared with the investigators and will be managed according to the agreements between the participating institutions and with the researchers. Data Property belongs to Fondazione Policlinico Universitario Campus Bio-Medico. The personnel involved in this study will have access to all data. In agreement with the ICH-GCP, the principal investigator of the study agrees to produce a report on the study, share all the data collected as described in the Protocol, and ensure that the data are reported responsibly and consistently.
  The transmission or dissemination of data through scientific publications and/or presentations in congresses, conferences, seminars, and participation in multicenter studies will take place exclusively following a purely statistical processing of the same, or in any case, in an anonymous form.

REFERENCES:
- [Derived] Spallone G, Mancini L, Carnevale A, Campi S, Schena E, D'Hooghe P, Hirschmann MT, Papalia R, Longo UG. Joint modeling and marker set selection significantly influence functional biomechanics in end-stage knee osteoarthritis: evidence from the sit-to-stand task. Front Bioeng Biotechnol. 2025 Oct 13;13:1677244. doi: 10.3389/fbioe.2025.1677244. eCollection 2025. PMID 41158195